CLINICAL TRIAL: NCT05157074
Title: Drum-PD/HD: The Impact of Group Drum-Based Music Therapy Intervention on Quality of Life and Motor Symptoms in Parkinson's Disease and Huntington's Disease
Brief Title: Group Drum-Based Music Therapy Intervention for Parkinson's Disease/Huntington's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00147450
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Huntington Disease
Keywords: group drumming; music therapy; motor function; quality of life; cognition; social and emotion; caregiver burden
MeSH Terms: conditions — Parkinson Disease; Huntington Disease; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Participants were assigned based on diagnosis, into two intervention groups 1) patients diagnosed with Parkinson's disease and the participant's study partners, 2) patients diagnosed with Huntington's disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Disease (PD) Group (Experimental): Participants with PD and their caregivers receive group drum classes twice a week for 12 weeks (24 lessons).
  Interventions: Behavioral: Group Drumming Music Therapy
- Huntington's Disease (HD) Group (Experimental): Participants with HD and their caregivers receive group drum classes twice a week for 12 weeks (24 lessons).
  Interventions: Behavioral: Group Drumming Music Therapy

INTERVENTIONS:
Behavioral: Group Drumming Music Therapy — All 24 Armstrong Rhythm Cycle™ sessions is conducted in a circle to ensure maximum line of sight for each participant. A variety of diverse percussion instruments ranging from hand drums, stick drums, shakers, and rhythm sticks are available as well as adaptive measures to address limited physical functioning. Instrument choice is dependent on ease of use for the level of the physical ability, skill development needs, and personal choice. Participants are informed that the participants free to use the same instrument for the duration of each session or to switch instruments at any time.
  Utilizing the five components of The Armstrong Rhythm Method, this protocol guides participants through three phases to achieve rhythmic skill development and group cohesion for therapeutic benefit.

SUMMARY:
Participants in this study (18-89 years) with Parkinson's disease or Huntington's disease receive drum classes twice a week for 12 weeks (24 lessons). All participants also participate in study visits for assessments before the beginning of the study, at the 6 week mark, at the 12 week mark and at the 18 week mark so that the investigators can assess the short and long term effects of drum classes on hand dexterity, upper extremity function and well-being.

DETAILED DESCRIPTION:
There has been evidence that rhythm-based music therapy interventions may improve motor outcomes for patients with Parkinson's disease and Huntington's disease, as well as quality of life for both patients and the patients' caregivers. DRUM-PD, a pilot study investigating the impact of West African drumming on quality of life, symptoms, motor findings, cognition, and mood in Parkinson's disease, found trends toward improvement in walking from baseline to 12 weeks and improved quality of life for patients who completed the 6 week drumming intervention. Building on this research, the investigators plan to evaluate the impact of a 12-week, twice weekly rhythm-based music therapy intervention called The Armstrong Rhythm Cycle℠, implemented by a board-certified music therapist. The investigators hypothesize that participation in 24 bi-weekly, hour-long music therapy drumming sessions will result in improved motor functioning for patients and better quality of life for patients and the patients' caregivers as compared to baseline before the intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients with Parkinson's Disease (PD) and Huntington's Disease (HD)

* Ability to give written consent
* Age 18-90
* Clinical diagnosis of probable of clinically established Parkinson disease; or Huntington disease confirmed by genetic testing (greater than or equal to 36 CAG repeats)
* Ability to move hands, wrists and arms safely for instrument play
* Presence of study partner who is available for all drum lessons and study assessments

Study Partners:

* Ability to give written consent
* Ability to give written consent
* Age 18-90
* Ability to move hands, wrists and arms safely for instrument play

Exclusion Criteria:

* PD: Hoehn & Yahr Stage 5 disease; Schwab & England score 40% or lower
* HD: Total Functional Capacity scores between 5 and 13 inclusive
* Co-morbid diagnosis (broken bones, sprains, severe arthritis, conditions involving paresis) in the judgement of the patient's treating physician that may preclude participant's full ability to participate in the intervention group.
* MoCA scores <17
* Active psychosis or other condition affecting the participants' ability to safely cooperate with study procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Changes in score on anxiety level as assessed by Neuro-QoL (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Neuro-QoL is a set of self-report measures that assess the health-related quality of life (HRQOL) of adults and with neurological disorders including PD and HD. For anxiety domain, unpleasant thoughts and/or feelings related to fear (e.g., fearfulness, feelings of panic), helplessness, worry and hyperarousal (e.g., tension, nervousness, restlessness) are measured.
  All Neuro-QoL items employ five response options (e.g., 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much)
  *High scores indicate worse (undesirable) self-reported health.
Changes in score on depression level as assessed by Neuro-QoL (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Neuro-QoL is a set of self-report measures that assess the health-related quality of life (HRQOL) of adults and with neurological disorders including PD and HD.
  For depression domain, experience of loss and feelings of hopelessness, negative mood (e.g., sadness, guilt), decrease in positive affect (e.g., loss of interest), information-processing deficits (e.g., problems in decision-making), negative views of the self (e.g., self-criticism, worthlessness), and negative social cognition (e.g., loneliness) are measured.
  All Neuro-QoL items employ five response options (e.g., 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much)
  *High scores indicate worse (undesirable) self-reported health.
Changes in score on upper extremity performance level as assessed by Neuro-QoL (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Neuro-QoL is a set of self-report measures that assess the health-related quality of life (HRQOL) of adults and with neurological disorders including PD and HD.
  For upper extremity domain, one's ability to carry out various activities involving digital, manual and reach-related functions, ranging from fine motor to self-care (activities of daily living) are measured.
  All Neuro-QoL items employ five response options (e.g., 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much)
  *High scores indicate better (desirable) self-reported health.
Changes in score on lower extremity performance level as assessed by Neuro-QoL (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Neuro-QoL is a set of self-report measures that assess the health-related quality of life (HRQOL) of adults and with neurological disorders including PD and HD.
  For lower extremity domain, one's ability to carry out various activities involving the trunk region and increasing degrees of bodily movement, ambulation, balance, or endurance are measured.
  All Neuro-QoL items employ five response options (e.g., 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much)
  *High scores indicate better (desirable) self-reported health.
Changes in score on ability to participate in social roles and activities as assessed by Neuro-QoL (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Neuro-QoL is a set of self-report measures that assess the health-related quality of life (HRQOL) of adults and with neurological disorders including PD and HD.
  For the ability to participate in social roles and activities domain, degree of involvement in one's usual social roles, activities and responsibilities, including work, family, friends, and leisure are measured.
  All Neuro-QoL items employ five response options (e.g., 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much)
  *High scores indicate better (desirable) self-reported health.
Changes in score on satisfaction with social roles and activities as assessed by Neuro-QoL (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Neuro-QoL is a set of self-report measures that assess the health-related quality of life (HRQOL) of adults and with neurological disorders including PD and HD.
  For the satisfaction with social roles and activities domain, satisfaction with involvement in one's usual social roles, activities and responsibilities, including work, family, friends, and leisure are measured.
  All Neuro-QoL items employ five response options (e.g., 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much)
  *High scores indicate better (desirable) self-reported health.
Changes in score on positive affect and well-being level as assessed by Neuro-QoL (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Neuro-QoL is a set of self-report measures that assess the health-related quality of life (HRQOL) of adults and with neurological disorders including PD and HD.
  For positive affect and well-being domain, aspects of a person's life that relate to a sense of well-being, life satisfaction or an overall sense of purpose and meaning are measured.
  All Neuro-QoL items employ five response options (e.g., 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much)
  *High scores indicate better (desirable) self-reported health.
Changes in score on burden level as assessed by the Zarit Burden Interview (ZBI) (study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The Zarit Burden Interview, a popular caregiver self-report measure used by many aging agencies, originated as a 29-item questionnaire. The 29-item instrument is included in Zarit et al., 1980. The revised version contains 22 items. This study used 22 items.
  It is scored as either (0) never, (1) rarely, (2) sometimes, (3) quite frequently, or (4) nearly always. Items are then summed and total scores are interpreted as follows: 0 to 21 little or no burden, 21 to 40 mild to moderate burden, 41 to 60 moderate to severe burden, and 61 to 88 severe burden.

SECONDARY OUTCOMES:
Changes in score on cognitive impairment level as assessed by the MoCA (patients) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Montreal Cognitive Assessment (MoCA) is a rapid cognitive screening test that assesses cognitive performance in multiple domains including visuo-spatial and executive functions, naming, memory, attention, language, abstraction, and orientation. Scores on the MoCA range from 0 to 30:
  > 26 = normal 18-25 = mild cognitive impairment 10-17 = moderate cognitive impairment <10 = severe cognitive impairment.
Change in score on depression level as assessed by the BDI-II (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  Beck-Depression inventory (BDI-II) measures characteristic attitudes and symptoms of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score for the Beck Depression Inventory-II (BDI-II).
  There is a four-point scale for each item ranging from 0 to 3. On two items (16 and 18) there are seven options to indicate either an increase or decrease of appetite and sleep. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Changes in score on the daily living level as assessed by Parkinson's Disease Questionnaire (PDQ-39) (patients) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. It also assesses the impact of Parkinson's on specific dimensions of functioning and wellbeing 5 point ordinal scoring system (lower scores reflect better QoL) 0 = never
  1. = occasionally
  2. = sometimes
  3. = often
  4. = always
Changes in score on patient health level as assessed by the short form (SF)-36 (patients and study partner) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
  The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Changes in score on apathy level as assessed by Apathy Evaluation Scale (patients) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The Apathy Evaluation Scale addresses characteristics of goal-directed behavior that reflect apathy including behavioral, cognitive, and emotional indicators (18 items).
  Items are scored on a 4-point Likert scale (not at all true, slightly true, somewhat true, very true).
  Score range: 18-72 (higher scores reflect more apathy)
Changes in score on non-motor aspects of experiences of daily living level as assessed by the Movement Disorder Society (MDS) sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (Part 1) (patients) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The MDS-UPDRS was developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. It includes a motor evaluation and characterizes the extent and burden of disease across various populations.
  Part 1 includes a total of 13 items.
  Items are scored on a 5-point Likert scale (normal, slight, mild, moderate, severe).
Changes in score on motor aspects of experiences of daily living level as assessed by the Movement Disorder Society (MDS) sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (Part 2) (patients) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The MDS-UPDRS was developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. It includes a motor evaluation and characterizes the extent and burden of disease across various populations.
  Part 2 includes a total of 13 items.
  Items are scored on a 5-point Likert scale (normal, slight, mild, moderate, severe).
Changes in score on motor examination level as assessed by the Movement Disorder Society (MDS) sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (Part 3) (patients) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The MDS-UPDRS was developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. It includes a motor evaluation and characterizes the extent and burden of disease across various populations.
  Part 3 includes a total of 18 items as well as dyskinesia related and Hoehn and Yahr stage items.
  Items are scored on a 5-point Likert scale (normal, slight, mild, moderate, severe).
Changes in score on motor complications level as assessed by the Movement Disorder Society (MDS) sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (Part 4) (patients) | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The MDS-UPDRS was developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. It includes a motor evaluation and characterizes the extent and burden of disease across various populations.
  Part 4 includes a total of 6 items.
  Items are scored on a 5-point Likert scale (normal, slight, mild, moderate, severe).
Changes in score on activities of daily living level as assessed by the Schwab and England scale | Baseline, 6 weeks, 12 weeks, and 18 weeks
  The Schwab and England ADL (Activities of Daily Living) scale is a method of assessing the capabilities of people with impaired mobility. The scale uses percentages to represent how much effort and dependence on others people need to complete daily chores. The rating may be given by a professional or by the person being tested.
  0% (fully dependent) to 100% completely independent)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Pantelyat, Principal Investigator — Department of Neurology, Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pantelyat A, Syres C, Reichwein S, Willis A. DRUM-PD: The use of a drum circle to improve the symptoms and signs of Parkinson's disease (PD). Mov Disord Clin Pract. 2016 May-Jun;3(3):243-249. doi: 10.1002/mdc3.12269. Epub 2015 Dec 21. PMID 27340683
- [Background] National Institute of Neurological Disorders and Stroke (NINDS). User Manual for the Quality of Life in Neurological Disorders (Neuro-QoL) Measures, Version 2.0, March 2015.
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Peto V, Jenkinson C, Fitzpatrick R, Greenhall R. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res. 1995 Jun;4(3):241-8. doi: 10.1007/BF02260863. PMID 7613534
- [Background] Beck AT, Steer RA, Brown GK. Manual for the beck depression inventory-II.1996
- [Background] Marin RS, Biedrzycki RC, Firinciogullari S. Reliability and validity of the Apathy Evaluation Scale. Psychiatry Res. 1991 Aug;38(2):143-62. doi: 10.1016/0165-1781(91)90040-v. PMID 1754629
- [Background] McRae C, Diem G, Vo A, O'Brien C, Seeberger L. Reliability of measurements of patient health status: a comparison of physician, patient, and caregiver ratings. Parkinsonism Relat Disord. 2002 Jan;8(3):187-92. doi: 10.1016/s1353-8020(01)00009-8. PMID 12039430
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914